CLINICAL TRIAL: NCT06284512
Title: Uveal Melanoma In Sonography and Color Fundus Photos - A Comparative Study
Brief Title: Uveal Melanoma - Comparative Study
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Told, MD, PhD, Medical University of Vienna
Other Study IDs: Uveal Melanoma 1942/2022
Record Dates: First submitted 2023-10-12; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uveal Melanoma: Patients with uveal melanoma will undergo a routine diagnostic imaging with color fundus photography and sonography.
  Interventions: Diagnostic Test: Sonography, color fundus photography

INTERVENTIONS:
Diagnostic Test: Sonography, color fundus photography — Patients will undergo routine diagnostic imaging (Sonography, color fundus photography)

SUMMARY:
The progress of uveal melanoma is typically monitored with sonography by experienced onco-ophthalmologists. However, there is evidence that twodimensional measurements in color fundus photography match precisely with sonography measurements. This study aims to compare sonography and color fundus photography measurements in order to evaluate the feasibility of monitoring of uveal melanoma with color fundus photography.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uveal melanoma

Exclusion Criteria:

* Inadequate or missing information on the clinical course in patient charts
* Imaging not feasible due to any reason.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uveal melanoma will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Largest Basal Diameter | 1 day
  Largest Basal Diameter will be measured on echography and color fundus photography

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Told, MD, PhD, Priv.-Doz., Principal Investigator — Deparment of Ophthalmology and Optometry
Locations (1):
- Medical University of Vienna, Department of Ophthalmology and Optometry, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No